CLINICAL TRIAL: NCT03448718
Title: Phase 2 Trial of Olaparib in Patients With Metastatic Urothelial Cancer Harboring DNA Damage Response Gene Alterations
Brief Title: Trial of Olaparib in Patients With Metastatic Urothelial Cancer Harboring DNA Damage Response Gene Alterations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Galsky (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Sponsor Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU15-262
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Urothelial Cancer
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olaparib Monotherapy (Experimental): The starting dose of olaparib tablets will be dependent on the subject's calculated creatinine clearance (CrCl). Subjects with a CrCl of ≥ 40 mL/min will start at a dose of olaparib tablets of 300 mg twice a day. Subjects with a CrCl of > 30 to < 40 mL/min will start at a dose of olaparib tablets 200 mg twice a day.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — 1 cycle = 28 days. Subject's with calculated creatinine clearance (CrCl) of ≥ 40 mL/min will start at a dose of olaparib tablets of 300 mg twice a day. Subjects with a CrCl of > 30 to < 40 mL/min will start at a dose of olaparib tablets 200 mg twice a day.
  Other Names: Lynparza

SUMMARY:
This is a single arm open label multi-institutional phase II trial of olaparib monotherapy in subjects with metastatic urothelial cancer harboring somatic DNA damage response (DDR) alterations. The primary objective of the study is to estimate the objective response rate (per RECIST 1.1) to treatment with olaparib.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of ≤ 1 within 14 days prior to registration. Cisplatin-ineligible chemotherapy-naïve subjects (see inclusion criteria #8) may have an ECOG Performance Status of ≤ 2.
* Histological or cytological evidence/confirmation of urothelial cancer.
* Metastatic and/or unresectable (cT4b) urothelial cancer.
* Metastatic disease evaluable on imaging studies. Subjects may have measurable disease according to RECIST 1.1 or bone-only disease within 30 days prior to registration.

  * NOTE: Bone-only subjects are eligible if their disease can be documented/ evaluated by bone scans, CT or MRI. Their disease will be assessed using MD Anderson criteria.34
  * NOTE: Previously irradiated lesions are eligible as a target lesion only if there is documented progression of the lesion after irradiation.
* Somatic alteration considered pathogenic/likely pathogenic in one of the following DDR genes as determined by genomic sequencing performed in a Clinical Laboratory Improvement Amendments (CLIA) laboratory. Somatic alterations will include nonsense, frameshift, splice-site or missense mutations or homozygous deletions. Subjects with alterations in DDR genes not included in the list below will be considered on a case by case basis after discussion with the sponsor-investigator(s). Subjects with germline alterations in DDR genes will be considered on a case by case basis and will be reviewed by the sponsor-investigator(s). At least 6 subjects will have BRCA or ATM alterations.
* Nucleotide Excision Repair: ERCC2, ERCC3,ERCC4, ERCC5, ERCC6
* Homologous Recombination: BRCA1, RAD52, BRCA2, RAD54L, RAD50, NBN RAD51, MRE11A, RAD51B, RAD51D, RAD51C, CTIP
* DNA Sensor: ATM, ATR, MDC1, ATRX, CHEK1, CHEK2
* Fanconi Anemia Pathway: PALB2, FANCE, BRIP1, FANCF, FANCA, FANCG FANCB, BLM, FANCC, FANCD2
* Base Excision Repair: XRCC2, XRCC3, XRCC4, XRCC5, XRCC6
* Other: MUTYH, RECQL4, POLQ, POLE, WRN
* A subject with prior brain metastasis may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to study registration, have been off of corticosteroids for ≥ 2 weeks, and are asymptomatic
* Subjects must have progressed despite at least 1 prior line of treatment for metastatic and/or unresectable urothelial cancer. However, cisplatin-ineligible (defined by a calculated creatinine clearance of >30 but < 60 mL/min OR CTCAE v4 Grade ≥ 2 audiometric hearing loss OR CTCAE v4 Grade ≥ 2 peripheral neuropathy OR ECOG PS = 2), and chemotherapy-naïve subjects are also eligible.
* Prior cancer treatment (systemic therapy or radiation therapy) must be completed at least 3 weeks prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to Grade ≤ 1 or baseline.
* Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 28 days prior to registration.

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Platelets ≥ 100 x 109/L
  * Calculated creatinine clearance ≥ 30 mL/min
  * Bilirubin ≤ 1.5 × upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN (or ≤ 5 × ULN if liver metastases)
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN (or ≤ 5 × ULN if liver metastases)
* Female subjects must be postmenopausal or there must be evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.
* Females of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of highly effective methods of contraception from the time of informed consent until 90 days after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method. Males must be willing to abstain from heterosexual activity or to use 2 forms of highly effective methods of contraception from the time of informed consent until 90 days after treatment discontinuation.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study
* 15. All subjects must have adequate archival tissue available prior to registration (i.e., at least 15 unstained slides or paraffin block). Archival tissue should represent invasive or metastatic urothelial cancer with a preference for metastatic tissue if available. Archival tissue should be identified at screening and shipped by C1D1. Subjects without adequate tissue may be considered on a case by case basis after discussion with the sponsor-investigator.

Exclusion Criteria

* Active infection requiring systemic therapy.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Known additional malignancy that is active and/or progressive requiring treatment; subjects with other malignancies that have been definitively treated and who have been rendered disease free will be eligible.
* Prior treatment with a PARP inhibitor, including olaparib.
* Treatment with any investigational drug within 30 days prior to registration.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Subjects with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
* Major surgery within 2 weeks of starting study treatment and subjects must have recovered from any effects of any major surgery.
* Subjects considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan, history of pneumonitis, or any psychiatric disorder that prohibits obtaining informed consent.
* Subjects unable to swallow orally administered medication and subjects with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Immunocompromised subjects, e.g., subjects who are known to be serologically positive for human immunodeficiency virus (HIV).
* Subjects with a known hypersensitivity to olaparib or any of the excipients of the product.
* Subjects with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
* Previous allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, MD, Principal Investigator — Mt Sinai School of Medicine
Locations (7):
- United States (7):
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Center (Wyane State University), Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt-Ingran Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olaparib Monotherapy
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Olaparib Monotherapy
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 66 [45 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Prior Systemic Therapies [Median (Full Range); unit: Lines of therapy] | 2 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  ORR is defined as the proportion of all subjects with confirmed PR or CR according to RECIST 1.1.
Time Frame: Up to a maximum of 17 months
Population: Out of 19 patients, four subjects were not evaluable for best response.
Measure: Number; unit: Percentage of participants
Arm/Group | Olaparib Monotherapy
Number analyzed (Participants) | 15
Percentage of participants | 0

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. PFS is defined as time from registration until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: Time of treatment start until the criteria for disease progression or death. Up to a maximum of 17 months.
Measure: Median (Full Range); unit: Months
Arm/Group | Olaparib Monotherapy
Number analyzed (Participants) | 19
Months | 1.9 [0.8 to 16.1]

3. Other Pre Specified Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from treatment start until death or date of last contact.
Time Frame: Time of treatment start until death or date of last contact, up to a maximum of 23 months.
Measure: Median (Full Range); unit: Months
Arm/Group | Olaparib Monotherapy
Number analyzed (Participants) | 19
Months | 9.5 [1.5 to 22.1]

4. Other Pre Specified Outcome: Adverse Events
Description: Number of participants with treatment related adverse events are reported by CTCAEv4 term and grade.
Time Frame: AE had been recorded from time of signed informed consent until 30 days after discontinuation of study drug(s) or until a new anti-cancer treatment starts, whichever occurs first, up to a maximum of 18 months.
Measure: Number; unit: Participants
Arm/Group | Olaparib Monotherapy
Number analyzed (Participants) | 19
Participants
  WBC count decreased | 1
  Lymphocyte count decreased | 2
  Neutrophil count decreased | 2
  Platelet count decreased | 3
  Anemia | 5
  Fatigue | 4
  Fever | 1
  Dizziness | 1
  Anorexia | 2
  Myalgia | 1
  Nausea | 4
  Vomiting | 3
  Diarrhea | 2
  Constipation | 1
  Abdominal pain | 1
  Allergic reaction | 1
  Confusion | 1
  Papulopustular rash | 1
  Skin disorders, other | 1
  Sore throat | 1
  Chronic kidney disease | 1
  Creatinine increased | 2

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 23 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 18 months.
Arm/Group | Olaparib Monotherapy
All-Cause Mortality (participants affected / at risk) | 13/19
Serious Adverse Events (participants affected / at risk) | 11/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib Monotherapy (N=19)
CONFUSION (Psychiatric disorders) | 1 (1)
CREATININE INCREASED (Investigations) | 1 (1)
EDEMA CEREBRAL (Nervous system disorders) | 1 (1)
FEVER (General disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (2)
LUNG INFECTION (Infections and infestations) | 2 (2)
PAIN (General disorders) | 1 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (2)
STROKE (Nervous system disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib Monotherapy (N=19)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (3)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (2)
ALLERGIC REACTION (Immune system disorders) | 1 (1)
ANAL MUCOSITIS (Gastrointestinal disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 10 (24)
ANOREXIA (Metabolism and nutrition disorders) | 4 (4)
ANXIETY (Psychiatric disorders) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
BLADDER SPASM (Renal and urinary disorders) | 2 (2)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 1 (3)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 2 (2)
CHOLESTEROL HIGH (Investigations) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 2 (2)
CONFUSION (Psychiatric disorders) | 1 (2)
CONSTIPATION (Gastrointestinal disorders) | 4 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CREATININE INCREASED (Investigations) | 7 (16)
DEPRESSION (Psychiatric disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 2 (2)
DIZZINESS (Nervous system disorders) | 2 (3)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
EDEMA LIMBS (General disorders) | 2 (3)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 1 (1)
FACIAL PAIN (General disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 2 (3)
FATIGUE (General disorders) | 10 (12)
FEVER (General disorders) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
GASTROPARESIS (Gastrointestinal disorders) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 3 (4)
HEADACHE (Nervous system disorders) | 1 (1)
HEMATOMA (Vascular disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 4 (4)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 3 (4)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 4 (6)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 4 (5)
HYPOTENSION (Vascular disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
LETHARGY (Nervous system disorders) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
LOCALIZED EDEMA (General disorders) | 1 (2)
LYMPHOCYTE COUNT DECREASED (Investigations) | 7 (10)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (7)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (2)
PAIN (General disorders) | 2 (5)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 5 (6)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 3 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 1 (3)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY (Reproductive system and breast disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (5)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT03448718/Prot_SAP_000.pdf